CLINICAL TRIAL: NCT00166283
Title: Improving New Learning in Multiple Sclerosis: A Randomized Clinical Trial
Brief Title: Improving New Learning and Memory in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ndcnih2004; R01HD045798 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Sclerosis
Keywords: memory; learning; Multiple Sclerosis; Cognition; treatment; therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): The experimental group will receive memory retraining exercises administered on a laptop computer twice a week for five weeks (10 training sessions).
  Interventions: Behavioral: memory retraining exercises
- placebo control group (Placebo Comparator): The placebo control group will receive placebo memory exercises administered on a laptop computer twice a week for five weeks (10 placebo control sessions).
  Interventions: Behavioral: placebo control memory exercises

INTERVENTIONS:
Behavioral: memory retraining exercises — Memory retraining exercises will be administered on a laptop computer twice a week for five weeks (10 training sessions).
  Arms: experimental group
Behavioral: placebo control memory exercises — Placebo control memory exercises will be administered on a laptop computer twice a week for five weeks (10 training sessions).
  Arms: placebo control group

SUMMARY:
The current study is a double-blind, placebo-control randomized clinical trial examining the efficacy of memory retraining in Multiple Sclerosis (MS). Impairment in higher level cognitive processing, such as new learning and memory, is one of the most common deficits in individuals with MS and such deficits have been shown to exert significant negative impact on multiple aspects of everyday life, including occupational and social functioning. Despite these findings, few studies have attempted to treat these cognitive deficits in order to improve the everyday functioning of individuals with MS. Through a small randomized clinical trial, we found that individuals with MS with documented memory impairment show a significant improvement in their memory performance following a treatment protocol designed to facilitate learning. The current proposal will replicate this finding and further evaluate (a) the impact of the treatment on everyday functioning, (b) the long term efficacy of the treatment and (c) the utility of booster sessions in facilitating long-term treatment effects. We will randomly assign individuals with MS, with documented impairment in new learning abilities, to a memory retraining group or a placebo control group. Both groups will undergo baseline, immediate and long-term follow-up assessment consisting of: (1) a traditional neuropsychological battery and (2) an assessment of global functioning examining the impact of the treatment on daily activities. This design will allow us to evaluate the efficacy of this particular memory retraining technique in an MS population through the assessment of cognitive function via a standard evaluation. In addition, we will be able to draw conclusions regarding the impact of this particular memory remediation program on everyday life from questionnaires completed by the participant and a significant other. Optional enrollment in pre- post neuroimaging will also allow us to look at changes in the brain.

DETAILED DESCRIPTION:
Impairments in higher level cognitive processing, such as new learning and memory, are among the most common deficits in individuals with Multiple Sclerosis (MS) and such deficits have been shown to exert significant negative impact on multiple aspects of everyday life, including occupational and social functioning. Despite these findings, few studies have attempted to remediate these cognitive deficits in order to improve the everyday functioning of individuals with MS. While limited research addressing the efficacy of memory retraining in MS does exist, this research has been marred by significant methodological flaws. Specifically, the only existing study of memory retraining in MS to utilize: (1) a randomized clinical trial and (2) an objective outcome assessment is our pilot research carried out at Kessler Medical Rehabilitation Research and Education Corporation (KMRREC).

"The Advisory Board recommends that NCMRR initiate and coordinate studies of the effectiveness of medical rehabilitation interventions…using new and precise quantitative measurements of impairment, including functional and societal limitations and disability, with particular emphasis on disability and societal limitations." The current proposal directly addresses this recommendation of the NCMRR Advisory Board. It is designed to (1) replicate our pilot study with larger sample sizes (2) expand our assessment measures to better assess individuals with mild cognitive impairments, thus testing the effectiveness of the intervention within this important subpopulation (3) assess the effectiveness of the intervention utilizing more global measures of everyday life, including an objective measure (the Rivermead Behavioral Memory Test), which has preliminary support through our pilot study, as well as additional questionnaires to be completed by both the participant and a significant other (4) evaluate the long-term effects of the treatment protocol and (5) examine the utility of booster sessions to facilitate long-term treatment effects.

To meet these study objectives, we will conduct a double-blind, placebo-controlled, randomized clinical trial, applying a memory rehabilitation technique to a large sample of MS participants. This protocol has been well-validated with other neurological populations and preliminary evidence in support of its use in MS now exists. Individuals with MS, with documented impairment in memory and new learning, will be randomly assigned to either a memory retraining group or a placebo control group. Outcome will be measured through several mechanisms: (1) a traditional neuropsychological (NP) battery and (2) an assessment of global functioning (AGF) examining the impact of the treatment on daily activities. Both groups will undergo baseline, immediate follow-up, and long-term follow-up assessments consisting of a traditional NP evaluation, which examines objective performance on well-validated measures of cognitive function, and an AGF, which includes self-report measures of memory abilities, self-efficacy, quality of life, and occupational functioning. In this way, we will be able to objectively evaluate the presence or absence of changes in memory performance through a NP assessment, while also evaluating the impact of this treatment protocol on an individual's everyday life through the AGF. While most studies evaluating the efficacy of cognitive retraining usually employ a pre-training and post-training evaluation, such evaluations have been criticized for their lack of ecological validity. The present design allows the assessment of the efficacy of this particular memory retraining technique within an MS population using traditional measures, as well as the assessment of the impact that such a rehabilitation technique has on everyday life. In addition, we will include a 6-month follow-up assessment to measure the long-term impact of this treatment on objective cognitive functioning, through a NP assessment, and everyday life, through an AGF. Finally, half of the participants in the experimental group will participate in monthly "booster sessions" following the completion of treatment and we will evaluate the impact of these sessions on the maintenance of treatment effects over time. A subset of the sample will also complete pre and post neuroimaging to evaluate changes in cerebral activation.

Many studies have shown that new learning is a key problem in MS. In addition, a small pilot study, funded by the National Multiple Sclerosis Society (NMSS) and administered by the current PI, tested this memory retraining protocol in an MS population. Results showed that when these deficits in new learning are treated, a significant improvement is noted in memory performance. However, the impact of the memory retraining protocol on everyday functioning remains unclear. The documentation of the efficacy of memory retraining in MS, particularly on everyday functioning, could have a significant impact on symptom management and quality of life in the lives of persons with MS. As such, specific aims of the current research protocol are as follows.

Aim 1. This study will objectively evaluate the clinical utility of a memory retraining protocol to improve performance on objective tests of new learning and memory in a large sample of individuals with MS with documented deficits in this area. This protocol has been previously utilized in a traumatic brain injury (TBI) population and a small pilot sample of individuals with MS, yielding promising data. NCMRR states that research analyzing existing rehabilitation techniques, empirically assessing their validity, and providing justification to the consumer and practitioners is required for the advancement of the field of medical rehabilitation research and recognizes this as a high priority research area. Our study does precisely this.

Aim 2. We will increase the generalizability and real life application of assessment techniques by assessing outcome following cognitive retraining with more global measures of everyday life. An objective measure of everyday functioning will be included, as well as numerous subjective measures of everyday functioning, which will be gathered via established self-report instruments, as well as ratings by a significant other.

Aim 3. This study will also assess the efficacy of this memory retraining protocol in a mildly impaired MS group, which has not been properly tested previously. Due to measurement ceiling effects in our pilot study, the utility of this technique to improve new learning and memory abilities in individuals with mild deficits has not yet been determined. The current study improves upon the measurement techniques used in the pilot study.

Aim 4: This study will evaluate the long-term efficacy of this memory retraining protocol through the inclusion of a 6-month follow-up assessment. Many cognitive remediation studies in the literature examine the efficacy of the treatment immediately following program completion. However, given the time, expense, and labor involved in such intensive treatment, it is important to demonstrate the long-term efficacy of such a program. The current study therefore goes beyond the typical protocol length to evaluate the long-term impact such treatment will have on objective testing and on an individual's daily life.

Aim 5: Booster sessions have been used to maximize the long term benefit of cognitive retraining in other patient populations. However, the utility of booster sessions has never been investigated in MS. An additional question we will address in the current treatment study is the impact of "booster sessions" following the completion of the treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* English as primary language
* diagnosis of multiple sclerosis

Exclusion Criteria:

* ages less than 30 or greater than 70
* Most recent exacerbation within one month
* Other Neurological History: head injury, stroke, seizures, or any other significant neurological history will not be included in the study
* Medications: persons on steroids, benzodiazepines, and/or neuroleptics will not be included
* Individuals with an active diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder I or II will be excluded from the study.
* Poor Visual Acuity (corrected vision in worse eye < 20/60), diplopia, or nystagmus
* Inability to understand directions and following one, two, and three step commands
* Intact New Learning and Memory: Only individuals that show impaired performance on a memory test will be included in the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Scores on memory tests | Three points in time: pre-treatment, immediately following treatment and 6 months after treatment is completed

SECONDARY OUTCOMES:
Reports of emotional functioning, memory functioning, quality of life and neuroimaging. | Three points in time: pre-treatment, immediately following treatment and 6 months after treatment is completed

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D Chiaravalloti, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation Research Center, West Orange, New Jersey, United States